CLINICAL TRIAL: NCT02760277
Title: A Phase II Open-label, Multicenter Extension Study to Assess the Long-term Safety and Efficacy of Vamorolone in Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: An Extension Study to Assess Vamorolone in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ReveraGen BioPharma, Inc. (Industry)
Collaborators: University of Pittsburgh (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Cooperative International Neuromuscular Research Group (Network); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VBP15-003; 1R44NS095423-01 (NIH); 1U34AR068616-01 (NIH)
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; vamorolone
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — VBP15 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level Group 1 (Experimental): Participants enrolled in Dose Level Group 1 will receive vamorolone 0.25 mg/kg/day.
  Interventions: Drug: Vamorolone 0.25 mg/day/day
- Dose Level Group 2 (Experimental): Participants enrolled in Dose Level Group 2 will receive vamorolone 0.75 mg/kg/day.
  Interventions: Drug: Vamorolone 0.75 mg/day/day
- Dose Level Group 3 (Experimental): Participants enrolled in Dose Level Group 3 will receive vamorolone 2.0 mg/kg/day.
  Interventions: Drug: Vamorolone 2.0 mg/day/day
- Dose Level Group 4 (Experimental): Participants enrolled in Dose Level Group 4 will receive vamorolone 6.0 mg/kg/day.
  Interventions: Drug: Vamorolone 6.0 mg/day/day

INTERVENTIONS:
Drug: Vamorolone 0.25 mg/day/day — Oral administration of 0.25 mg/kg/day daily for 24 weeks.
  Other Names: VBP15
  Arms: Dose Level Group 1
Drug: Vamorolone 0.75 mg/day/day — Oral administration of 0.75 mg/kg/day daily for 24 weeks.
  Other Names: VBP15
  Arms: Dose Level Group 2
Drug: Vamorolone 2.0 mg/day/day — Oral administration of 2.0 mg/kg/day daily for 24 weeks.
  Other Names: VBP15
  Arms: Dose Level Group 3
Drug: Vamorolone 6.0 mg/day/day — Oral administration of 6.0 mg/kg/day daily for 24 weeks.
  Other Names: VBP15
  Arms: Dose Level Group 4

SUMMARY:
The main purposes of this study are to see if it is safe to use a new medication called vamorolone for more than two weeks in children with Duchenne muscular dystrophy (DMD), to see if vamorolone works for the treatment for DMD, and to see how any potential side effects compare to those seen in boys using steroids.

DETAILED DESCRIPTION:
This study will evaluate if it is safe to use a new medication called vamorolone for more than two weeks in children with DMD, if boys with DMD who take the study medication have improved muscle function compared to boys with DMD in other studies who did not take any type of steroid, and to see if boys with DMD who take the study medication gain less weight compared to boys with DMD in a prior study who took another type of steroid called prednisone. Enrolled participants will take the study medication for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant's parent or legal guardian has provided written informed consent/HIPAA authorization prior to any extension study-specific procedures;
2. Participant has previously completed study VBP15-002 up to and including the Week 4 Follow-up assessments within 8 weeks prior to enrollment; and
3. Participant and parent/guardian are willing and able to comply with scheduled visits, study drug administration plan, and study procedures.

Exclusion Criteria:

1. Participant had a serious or severe adverse event in study VBP15-002 that, in the opinion of the Investigator, was probably or definitely related to vamorolone use and precludes safe use of vamorolone for the subject in this study;
2. Participant has current or history of major renal or hepatic impairment, diabetes mellitus or immunosuppression;
3. Participant has current or history of chronic systemic fungal or viral infections;
4. Participant has used mineralocorticoid receptor agents, such as spironolactone, eplerenone, canrenone (canrenoate potassium), prorenone (prorenoate potassium), mexrenone (mexrenoate potassium) within 4 weeks prior to the first dose of study medication;
5. Participant has evidence of symptomatic cardiomyopathy. [Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary];
6. Participant is currently being treated or has received previous treatment with oral glucocorticoids or other immunosuppressive agents. [Notes: Past transient use of oral glucocorticoids or other oral immunosuppressive agents for no longer than 3 months cumulative, with last use at least 3 months prior to first dose of study medication, will be considered for eligibility on a case-by-case basis. Inhaled and/or topical corticosteroids prescribed for an indication other than DMD are permitted but must be administered at stable dose for at least 3 months prior to study drug administration];
7. Subject has used idebenone within 4 weeks prior to the first dose of study medication;
8. Participant has an allergy or hypersensitivity to the study medication or to any of its constituents;
9. Participant has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the Investigator;
10. Participant has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator; or
11. Participant is currently taking any investigational drug, or has taken any investigational drug other than vamorolone within 3 months prior to the start of study treatment.

Note: Participants may be re-evaluated if ineligible due to a transient condition which would prevent the subject from participating

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Clemens, MD, Study Chair — University of Pittsburgh
Locations (12):
- United States (6):
  - University of California Davis, Davis, California
  - University of Florida, Gainesville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (2):
  - Royal Children's Hospital, Melbourne
  - Sydney Children's Hospital, Westmead
- Alberta Children's Hospital, Calgary, Alberta, Canada
- Schneider Children's Medical Center, Petah Tikva, Israel
- Queen Silvia Children's Hospital, Gothenburg, Sweden
- Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Hoffman E, Gaglianone S, Ketema R, Tu W, Peay H, Clemens P, Dang U, Conklin L. Return of participant-level clinical trial results to participants: pilot of a simplified centralised approach. BMJ Open. 2024 Mar 23;14(3):e080097. doi: 10.1136/bmjopen-2023-080097. PMID 38521535
- [Derived] Smith EC, Conklin LS, Hoffman EP, Clemens PR, Mah JK, Finkel RS, Guglieri M, Tulinius M, Nevo Y, Ryan MM, Webster R, Castro D, Kuntz NL, Kerchner L, Morgenroth LP, Arrieta A, Shimony M, Jaros M, Shale P, Gordish-Dressman H, Hagerty L, Dang UJ, Damsker JM, Schwartz BD, Mengle-Gaw LJ, McDonald CM; CINRG VBP15 and DNHS Investigators. Efficacy and safety of vamorolone in Duchenne muscular dystrophy: An 18-month interim analysis of a non-randomized open-label extension study. PLoS Med. 2020 Sep 21;17(9):e1003222. doi: 10.1371/journal.pmed.1003222. eCollection 2020 Sep. PMID 32956407
- [Derived] Li X, Conklin LS, van den Anker J, Hoffman EP, Clemens PR, Jusko WJ. Exposure-Response Analysis of Vamorolone (VBP15) in Boys With Duchenne Muscular Dystrophy. J Clin Pharmacol. 2020 Oct;60(10):1385-1396. doi: 10.1002/jcph.1632. Epub 2020 May 20. PMID 32434278

RESULTS

PARTICIPANT FLOW:
Period: Vamorolone 0.25 mg/kg/Day
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Started | 12 | 0 | 0 | 0
Completed | 12 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: 0.75 mg/kg/Day
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Started | 0 | 12 | 0 | 0
Completed | 0 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: 2.0 mg/kg/Day
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Started | 0 | 0 | 12 | 0
Completed | 0 | 0 | 12 | 0
Not Completed | 0 | 0 | 0 | 0
Period: 6.0 mg/kg/Day
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Started | 0 | 0 | 0 | 12
Completed | 0 | 0 | 0 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who receive at least one dose of vamorolone study medication in the extension study will be included in the Safety Population. The Safety Population is the primary analysis population for safety assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 5.2 (1.03) | 4.8 (0.83) | 4.7 (0.89) | 4.8 (0.75) | 4.9 (0.87)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12 | 12 | 12 | 12 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 12 | 11 | 12 | 9 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 11 | 10 | 12 | 12 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 0 | 2 | 2 | 7
  Sweden | 0 | 4 | 0 | 0 | 4
  United States | 9 | 3 | 2 | 6 | 20
  United Kingdom | 0 | 0 | 4 | 2 | 6
  Israel | 0 | 3 | 2 | 0 | 5
  Australia | 0 | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as Assessed by CTCAE Version 4.03
Description: Treatment-emergent adverse events (TEAEs) are defined as any adverse event or worsening of an existing conditions after initiation of the investigational product and through the subject's last study visit (study completion or early termination). Serious adverse events were recorded for up to 30 days after the final administration of study drug; To evaluate the long-term safety and tolerability of vamorolone, administered orally at daily doses up to 6.0 mg/kg/day over a 24- week Treatment Period, in boys ages 4-7 years with DMD.
Time Frame: 24 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
participants
  Subjects with Any TEAE | 10 | 10 | 11 | 11
  Subjects with Any Drug Related TEAE | 1 | 2 | 4 | 5
  Subjects with Any CTCAE Grade 3 or Higher TEAE | 0 | 0 | 0 | 2
  Discontinuation of Study Drug due to TEAE | 0 | 0 | 0 | 0
  Subjects with Any Serious TEAE | 0 | 1 | 0 | 2
  Death | 0 | 0 | 0 | 0

2. Primary Outcome: Total Number of Adverse Events as Assessed by CTCAE Version 4.03
Description: as for outcome 1
Time Frame: 24 weeks
Population: as for baseline characteristics
Measure: Number; unit: Events
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
Events
  Total Number of AEs | 48 | 44 | 54 | 73
  Total Number of TEAEs | 48 | 44 | 54 | 72

3. Primary Outcome: Muscle Function Measured by Time to Stand Test (TTSTAND)- Velocity
Description: To compare the efficacy, as measured by the Time to Stand Test (TTSTAND), of vamorolone administered orally at daily doses up to 6.0 mg/kg over a 24-week Treatment Period vs. untreated DMD historical controls in boys ages 4-7 years with DMD
Time Frame: 002 Baseline, 003 Baseline, 003 Week 12, Week 24 (Note: 002 Baseline is from VBP15-002 4 week study (NCT02760264), previous to VBP15-003)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Rises/Second
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
Rises/Second
  002 Baseline | 0.18 (0.065) | 0.24 (0.090) | 0.22 (0.082) | 0.19 (0.056)
  003 Baseline | 0.15 (0.045) | 0.22 (0.077) | 0.24 (0.078) | 0.22 (0.070)
  003 Week 12: number analyzed (Participants) | 11 | 12 | 12 | 11
  003 Week 12 | 0.18 (0.072) | 0.23 (0.102) | 0.24 (0.089) | 0.22 (0.075)
  003 Week 12 Change from 002 Baseline: number analyzed (Participants) | 11 | 12 | 12 | 11
  003 Week 12 Change from 002 Baseline | -0.01 (0.061) | 0.00 (0.054) | 0.02 (0.066) | 0.02 (0.034)
  003 Week 24: number analyzed (Participants) | 10 | 12 | 12 | 11
  003 Week 24 | 0.18 (0.081) | 0.24 (0.114) | 0.26 (0.108) | 0.24 (0.086)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 10 | 12 | 12 | 11
  003 Week 24 Change from 002 Baseline | -0.01 (0.066) | 0.00 (0.062) | 0.05 (0.061) | 0.04 (0.045)

4. Primary Outcome: BMI Z-score
Description: Summary of BMI Z-score of Safety Population.
  Please note 0 is the mean. A negative result indicates a response that is many standard deviations below the mean, and a positive result indicates a response that is many standard deviations above the mean. In this case, the closer the group mean BMI Z-score is to 0 is more favorable.
Time Frame: 002 Baseline, 003 Week 12, Week 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
z score
  002 Baseline | 1.165 (0.6219) | 0.703 (1.0738) | 1.200 (0.5325) | 0.695 (0.7189)
  003 Week 12: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 | 1.103 (0.6457) | 0.494 (1.0680) | 1.261 (0.3981) | 1.011 (0.7034)
  003 Week 12 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 Change from 002 Baseline | -0.062 (0.2438) | -0.209 (0.4078) | 0.062 (0.3886) | 0.174 (0.5826)
  003 Week 24: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 24 | 1.004 (0.6381) | 0.493 (1.1696) | 1.242 (0.4596) | 1.330 (0.5857)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 24 Change from 002 Baseline | -0.161 (0.3234) | -0.210 (0.3629) | 0.043 (0.3849) | 0.493 (0.6363)

5. Secondary Outcome: Serum Pharmacodynamics Biomarkers Measured by Levels of HbA1c
Description: To investigate the effects of vamorolone, administered orally at daily doses up to 6.0 mg/kg over a 24-week Treatment Period vs. prednisone-treated historical controls, on serum pharmacodynamic (PD) biomarkers of safety (insulin resistance, adrenal axis suppression, and bone turnover). SomaScan aptamer panels testing 1,200 serum proteins were used to discover a candidate set of prednisone-responsive biomarkers, with a subset of these validating in a longitudinal sample set (individual DMD patients pre/post steroid treatment). These PD biomarkers were assigned to a safety panel or efficacy panel based on comparison to normal controls and information concerning the function of each protein.
Time Frame: 002 Baseline, 003 Week 8, 003 Week 16, 003 Week 24, 003 Week 26-29
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
% of HbA1c
  002 Baseline | 5.18 (0.260) | 5.22 (0.244) | 5.19 (0.124) | 5.23 (0.231)
  003 Week 8: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 8 | 5.18 (0.226) | 5.33 (0.250) | 5.28 (0.204) | 5.25 (0.216)
  003 Week 8 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 8 Change from 002 Baseline | 0.00 (0.128) | 0.12 (0.153) | 0.09 (0.198) | 0.00 (0.100)
  003 Week 16: number analyzed (Participants) | 12 | 11 | 12 | 11
  003 Week 16 | 5.26 (0.239) | 5.35 (0.238) | 5.26 (0.156) | 5.31 (0.270)
  003 Week 16 Change from 002 Baseline: number analyzed (Participants) | 12 | 11 | 12 | 11
  003 Week 16 Change from 002 Baseline | 0.08 (0.204) | 0.14 (0.225) | 0.07 (0.130) | 0.05 (0.113)
  003 Week 24: number analyzed (Participants) | 8 | 12 | 12 | 11
  003 Week 24 | 5.15 (0.302) | 5.22 (0.221) | 5.13 (0.160) | 5.24 (0.254)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 8 | 12 | 12 | 11
  003 Week 24 Change from 002 Baseline | -0.10 (0.220) | 0.00 (0.186) | -0.07 (0.130) | -0.02 (0.154)
  003 Week 26-29: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 | 5.07 (0.208) |  |  |
  003 Week 26-29 Change from 002 Baseline: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 Change from 002 Baseline | -0.07 (0.208) |  |  |

6. Secondary Outcome: Serum Pharmacodynamics Biomarkers Measured by Levels of HbA1c
Description: as for outcome 5
Time Frame: 002 Baseline, 003 Week 8, 003 Week 16, 003 Week 24, 003 Week 26-29
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
% change
  003 Week 8 % Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 8 % Change from 002 Baseline | 0.06 (2.470) | 2.28 (3.008) | 1.79 (3.864) | 0.02 (1.927)
  003 Week 16 % Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 16 % Change from 002 Baseline | 1.70 (3.989) | 2.72 (4.457) | 1.30 (2.505) | 1.03 (2.14)
  003 Week 24 % Change from 002 Baseline: number analyzed (Participants) | 8 | 12 | 12 | 11
  003 Week 24 % Change from 002 Baseline | -1.89 (4.801) | 0.08 (3.629) | -1.27 (2.525) | -0.33 (2.895)
  003 Week 26-29 % Change from 002 Baseline: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 % Change from 002 Baseline | -1.25 (3.942) |  |  |

7. Secondary Outcome: Serum Pharmacodynamics Biomarkers Measured by Levels of ACTH
Description: as for outcome 5
Time Frame: 002 Baseline, 003 Baseline, 003 Week 8, 003 Week 16, 003 Week 24, 003 Week 26-29 (Note: 002 Baseline is from VBP15-002 4 week study (NCT02760264), previous to VBP15-003)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
pg/mL
  002 Baseline: number analyzed (Participants) | 12 | 11 | 12 | 12
  002 Baseline | 18.3 (2.96) | 18.0 (6.88) | 21.1 (6.13) | 19.3 (8.67)
  003 Baseline | 15.9 (4.52) | 18.6 (4.56) | 18.2 (5.29) | 18.4 (9.73)
  003 Week 8: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 8 | 13.0 (6.25) | 7.1 (5.84) | 7.8 (4.42) | 6.5 (5.23)
  003 Week 8 Change from 002 Baseline: number analyzed (Participants) | 12 | 11 | 12 | 11
  003 Week 8 Change from 002 Baseline | -5.3 (6.92) | -10.5 (9.32) | -13.3 (7.33) | -13.5 (7.84)
  003 Week 16: number analyzed (Participants) | 11 | 11 | 12 | 9
  003 Week 16 | 12.2 (4.93) | 9.0 (5.86) | 9.0 (14.18) | 9.0 (4.49)
  003 Week 16 Change from 002 Baseline: number analyzed (Participants) | 11 | 10 | 12 | 9
  003 Week 16 Change from 002 Baseline | -6.2 (6.34) | -9.1 (9.89) | -12.0 (15.42) | -12.2 (8.16)
  003 Week 24: number analyzed (Participants) | 8 | 12 | 12 | 10
  003 Week 24 | 19.8 (6.32) | 14.0 (3.88) | 15.7 (9.63) | 11.3 (7.52)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 8 | 11 | 12 | 10
  003 Week 24 Change from 002 Baseline | 0.6 (6.63) | -4.0 (5.48) | -5.4 (11.09) | -6.3 (7.78)
  003 Week 26-29: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 | 9.5 (7.26) |  |  |
  003 Week 26-29 Change from 002 Baseline: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 Change from 002 Baseline | -7.8 (4.19) |  |  |

8. Secondary Outcome: Serum Pharmacodynamics Biomarkers Measured by Levels of Fasting Glucose
Description: as for outcome 5
Time Frame: 002 Baseline, 003 Week 12, 003 Week 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
mg/dL
  002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 10
  002 Baseline | 87.5 (9.44) | 88.9 (18.71) | 89.3 (7.91) | 92.3 (8.19)
  003 Week 12: number analyzed (Participants) | 11 | 10 | 12 | 11
  003 Week 12 | 81.5 (5.61) | 81.7 (4.35) | 84.3 (8.13) | 86.5 (5.57)
  003 Week 12 Change from 002 Baseline: number analyzed (Participants) | 11 | 10 | 12 | 10
  003 Week 12 Change from 002 Baseline | -6.8 (8.29) | -7.6 (19.22) | -5.1 (9.01) | -5.2 (9.21)
  003 Week 24: number analyzed (Participants) | 10 | 10 | 10 | 11
  003 Week 24 | 80.8 (6.56) | 80.8 (4.08) | 81.3 (7.94) | 84.6 (6.53)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 10 | 10 | 10 | 10
  003 Week 24 Change from 002 Baseline | -6.3 (11.97) | -9.0 (20.87) | -8.1 (10.28) | -7.8 (9.44)

9. Secondary Outcome: Serum Pharmacodynamics Biomarkers Measured by Levels of Fasting Insulin
Description: as for outcome 5
Time Frame: 002 Baseline, 003 Week 12, 003 Week 24
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
uIU/mL
  002 Baseline: number analyzed (Participants) | 11 | 8 | 12 | 12
  002 Baseline | 5.54 (3.651) | 3.09 (2.033) | 3.40 (1.548) | 3.96 (2.027)
  003 Week 12: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 | 4.17 (3.167) | 2.97 (1.669) | 3.89 (2.189) | 6.97 (3.526)
  003 Week 12 Change from 002 Baseline: number analyzed (Participants) | 11 | 8 | 12 | 11
  003 Week 12 Change from 002 Baseline | -1.13 (3.822) | -0.14 (1.756) | 0.49 (2.592) | 2.97 (2.277)
  003 Week 24: number analyzed (Participants) | 11 | 9 | 9 | 7
  003 Week 24 | 4.23 (2.560) | 3.12 (1.788) | 4.82 (3.393) | 7.21 (2.374)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 10 | 5 | 9 | 7
  003 Week 24 Change from 002 Baseline | -1.67 (4.478) | 0.34 (2.898) | 1.36 (3.262) | 3.26 (2.862)

10. Secondary Outcome: Serum Pharmacodynamics Biomarkers Measured by Levels of Osteocalcin
Description: as for outcome 5
Time Frame: as for outcome 7
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL
  002 Baseline | 37.94 (11.622) | 35.66 (6.800) | 41.17 (5.617) | 44.36 (5.979)
  003 Baseline | 39.20 (14.136) | 41.84 (8.552) | 47.91 (6.648) | 42.81 (10.851)
  003 Week 8: number analyzed (Participants) | 11 | 12 | 12 | 11
  003 Week 8 | 36.21 (10.374) | 41.78 (13.856) | 44.45 (7.439) | 41.55 (5.446)
  003 Week 8 Change from 002 Baseline: number analyzed (Participants) | 11 | 12 | 12 | 11
  003 Week 8 Change from 002 Baseline | -1.60 (8.849) | 6.13 (10.440) | 3.28 (8.325) | -2.01 (8.898)
  003 Week 16: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 16 | 39.01 (9.620) | 42.23 (9.393) | 44.60 (9.534) | 39.39 (6.972)
  003 Week 16 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 16 Change from 002 Baseline | 1.07 (9.916) | 6.57 (6.709) | 3.43 (10.718) | -4.17 (8.494)
  003 Week 24: number analyzed (Participants) | 7 | 12 | 12 | 10
  003 Week 24 | 38.80 (6.292) | 51.41 (11.265) | 51.98 (9.372) | 49.08 (7.771)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 7 | 12 | 12 | 10
  003 Week 24 Change from 002 Baseline | -1.34 (11.289) | 15.75 (10.211) | 10.81 (7.542) | 5.29 (7.858)
  003 Week 26-29: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 | 40.10 (18.729) |  |  |
  003 Week 26-29 Change from 002 Baseline: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 Change from 002 Baseline | -1.23 (17.943) |  |  |

11. Secondary Outcome: Serum Pharmacodynamics Biomarkers Measured by Levels of P1NP
Description: as for outcome 5
Time Frame: as for outcome 7
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL
  002 Baseline: number analyzed (Participants) | 12 | 11 | 12 | 12
  002 Baseline | 555.8 (184.72) | 480.7 (118.20) | 508.2 (94.36) | 511.5 (106.50)
  003 Baseline | 573.9 (251.02) | 489.3 (121.66) | 492.0 (81.92) | 566.3 (149.32)
  003 Week 8: number analyzed (Participants) | 11 | 12 | 12 | 11
  003 Week 8 | 511.6 (190.94) | 459.8 (101.93) | 485.2 (105.12) | 402.7 (70.46)
  003 Week 8 Change from 002 Baseline: number analyzed (Participants) | 11 | 11 | 12 | 11
  003 Week 8 Change from 002 Baseline | -20.3 (120.32) | -22.9 (128.79) | -23.0 (96.84) | -105.6 (121.07)
  003 Week 16: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 16 | 481.9 (159.93) | 431.8 (81.25) | 455.7 (99.50) | 488.5 (130.11)
  003 Week 16 Change from 002 Baseline: number analyzed (Participants) | 12 | 11 | 12 | 11
  003 Week 16 Change from 002 Baseline | -73.8 (109.31) | -42.4 (109.07) | -52.5 (104.05) | -19.8 (130.12)
  003 Week 24: number analyzed (Participants) | 8 | 12 | 12 | 10
  003 Week 24 | 457.1 (129.21) | 471.1 (121.10) | 565.5 (158.89) | 526.2 (130.18)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 8 | 11 | 12 | 10
  003 Week 24 Change from 002 Baseline | -30.8 (113.64) | 2.1 (165.16) | 57.3 (150.36) | 8.7 (88.95)
  003 Week 26-29: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 | 619.0 (379.07) |  |  |
  003 Week 26-29 Change from 002 Baseline: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 Change from 002 Baseline | -152.0 (331.46) |  |  |

12. Secondary Outcome: Serum Pharmacodynamics Biomarkers Measured by Levels of CTX
Description: as for outcome 5
Time Frame: 002 Baseline, 003 Baseline, 003 Week 8, 003 Week 16, Week 24, 003 Week 26-29 (Note: 002 Baseline is from VBP15-002 4 week study (NCT02760264), previous to VBP15-003)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
pg/mL
  002 Baseline: number analyzed (Participants) | 11 | 10 | 12 | 12
  002 Baseline | 871.0 (160.85) | 935.8 (286.50) | 936.8 (256.25) | 889.3 (186.68)
  003 Baseline | 915.9 (263.13) | 964.4 (319.26) | 949.8 (303.76) | 989.2 (216.29)
  003 Week 8: number analyzed (Participants) | 11 | 12 | 12 | 11
  003 Week 8 | 897.1 (365.45) | 933.3 (330.20) | 928.3 (333.11) | 825.5 (164.36)
  003 Week 8 Change from 002 Baseline: number analyzed (Participants) | 11 | 10 | 12 | 11
  003 Week 8 Change from 002 Baseline | 26.1 (368.76) | -31.6 (236.34) | -8.5 (248.82) | -59.6 (259.08)
  003 Week 16: number analyzed (Participants) | 12 | 12 | 12 | 10
  003 Week 16 | 885.4 (261.53) | 912.8 (305.08) | 939.8 (157.17) | 953.7 (199.53)
  003 Week 16 Change from 002 Baseline: number analyzed (Participants) | 11 | 10 | 12 | 10
  003 Week 16 Change from 002 Baseline | -2.6 (304.50) | -46.3 (321.06) | 3.0 (244.71) | 102.3 (230.44)
  003 Week 24: number analyzed (Participants) | 8 | 12 | 10 | 10
  003 Week 24 | 1109.3 (287.92) | 1235.6 (295.79) | 1248.7 (308.90) | 1237.0 (277.20)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 8 | 10 | 10 | 10
  003 Week 24 Change from 002 Baseline | 212.3 (318.86) | 295.6 (357.93) | 346.5 (327.16) | 321.4 (264.65)
  003 Week 26-29: number analyzed (Participants) | 3 | 0 | 0 | 0
  003 Week 26-29 | 1059.3 (536.26) |  |  |
  003 Week 26-29 Change from 002 Baseline: number analyzed (Participants) | 2 | 0 | 0 | 0
  003 Week 26-29 Change from 002 Baseline | 569.5 (28.99) |  |  |

13. Secondary Outcome: Muscle Strength, Mobility, and Functional Exercise Capacity as Measured by Time to Climb Test (TTCLIMB)- Velocity
Description: To investigate the effects of vamorolone, administered orally at daily doses up to 6.0 mg/kg over a 24-week Treatment Period, on muscle strength, mobility and functional exercise capacity vs. historical controls as measured by Time to Climb Test (TTCLIMB) in boys ages 4-7 years with DMD.
Time Frame: 002 Baseline, 003 Baseline, 003 Week 12, 003 Week 24 (Note: 002 Baseline is from VBP15-002 4 week study (NCT02760264), previous to VBP15-003)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: tasks/ second
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
tasks/ second
  002 Baseline | 0.20 (0.054) | 0.29 (0.147) | 0.29 (0.164) | 0.24 (0.086)
  003 Baseline | 0.20 (0.065) | 0.29 (0.168) | 0.31 (0.144) | 0.25 (0.082)
  003 Week 12: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 | 0.21 (0.064) | 0.34 (0.238) | 0.31 (0.157) | 0.26 (0.095)
  003 Week 12 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 Change from 002 Baseline | 0.01 (0.044) | 0.05 (0.115) | 0.02 (0.107) | 0.02 (0.051)
  003 Week 24: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 24 | 0.20 (0.071) | 0.30 (0.166) | 0.34 (0.148) | 0.29 (0.097)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 24 Change from 002 Baseline | 0.00 (0.076) | 0.01 (0.066) | 0.04 (0.090) | 0.05 (0.061)

14. Secondary Outcome: Muscle Strength, Mobility, and Functional Exercise Capacity as Measured by Time to Run/Walk 10 Meters Test (TTRW)- Velocity
Description: To investigate the effects of vamorolone, administered orally at daily doses up to 6.0 mg/kg over a 24-week Treatment Period, on muscle strength, mobility and functional exercise capacity vs. historical controls as measured by Time to Run/Walk Test (TTRW) in boys ages 4-7 years with DMD.
Time Frame: as for outcome 13
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: meters/ second
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
meters/ second
  002 Baseline | 1.60 (0.312) | 1.77 (0.367) | 1.84 (0.347) | 1.64 (0.279)
  003 Baseline | 1.57 (0.371) | 1.78 (0.414) | 1.86 (0.418) | 1.72 (0.295)
  003 Week 12: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 | 1.54 (0.306) | 1.77 (0.550) | 1.97 (0.503) | 1.88 (0.341)
  003 Week 12 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 Change from 002 Baseline | -0.06 (0.261) | 0.00 (0.307) | 0.13 (0.316) | 0.26 (0.297)
  003 Week 24: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 24 | 1.55 (0.384) | 1.84 (0.486) | 1.90 (0.321) | 1.89 (0.378)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 24 Change from 002 Baseline | -0.05 (0.311) | 0.06 (0.210) | 0.06 (0.210) | 0.27 (0.254)

15. Secondary Outcome: Muscle Strength, Mobility, and Functional Exercise Capacity as Measured by North Star Ambulatory Assessment (NSAA)
Description: To investigate the effects of vamorolone, administered orally at daily doses up to 6.0 mg/kg over a 24-week Treatment Period, on muscle strength, mobility and functional exercise capacity vs. historical controls as measured by North Star Ambulatory Assessment (NSAA) in boys ages 4-7 years with DMD. ***Total NSAA score is being reported. The score can range from 0 to 32. Higher scores (approaching 32) indicate a better outcome assessing functional mobility.
Time Frame: as for outcome 13
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
scores on a scale
  002 Baseline | 19.0 (5.13) | 20.5 (5.58) | 20.0 (4.95) | 19.7 (4.94)
  003 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Baseline | 20.1 (7.30) | 20.8 (5.66) | 21.7 (3.87) | 20.4 (4.01)
  003 Week 12: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 | 19.3 (5.60) | 21.2 (6.45) | 21.0 (5.13) | 20.4 (5.41)
  003 Week 12 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 12 Change from 002 Baseline | 0.3 (2.06) | 0.7 (2.71) | 1.0 (2.56) | 0.5 (2.38)
  003 Week 24: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 24 | 19.8 (7.09) | 21.6 (7.23) | 22.3 (3.80) | 22.3 (5.76)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  003 Week 24 Change from 002 Baseline | 0.8 (2.83) | 1.1 (2.94) | 2.3 (1.78) | 2.5 (2.62)

16. Secondary Outcome: Muscle Strength, Mobility, and Functional Exercise Capacity vs. Historical Controls as Measured by 6-minute Walk Test (6MWT) Meters
Description: To investigate the effects of vamorolone, administered orally at daily doses up to 6.0 mg/kg over a 24-week Treatment Period, on muscle strength, mobility and functional exercise capacity vs. historical controls as measured by 6-minute Walk Test (6MWT) in boys ages 4-7 years with DMD.
Time Frame: as for outcome 13
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
Meters
  002 Baseline: number analyzed (Participants) | 11 | 12 | 10 | 11
  002 Baseline | 316.2 (59.47) | 331.5 (52.76) | 353.9 (65.40) | 336.8 (63.18)
  003 Baseline: number analyzed (Participants) | 12 | 12 | 10 | 11
  003 Baseline | 294.3 (60.62) | 332.2 (56.83) | 341.1 (49.42) | 335.1 (80.13)
  003 Week 12: number analyzed (Participants) | 11 | 11 | 10 | 9
  003 Week 12 | 312.9 (60.93) | 358.7 (71.47) | 393.7 (59.72) | 369.9 (69.47)
  003 Week 12 Change from 002 Baseline: number analyzed (Participants) | 10 | 11 | 10 | 9
  003 Week 12 Change from 002 Baseline | 6.0 (28.81) | 20.8 (38.09) | 39.8 (35.61) | 27.6 (42.00)
  003 Week 24: number analyzed (Participants) | 10 | 12 | 10 | 10
  003 Week 24 | 306.2 (68.08) | 350.4 (64.23) | 383.1 (63.38) | 372.6 (69.12)
  003 Week 24 Change from 002 Baseline: number analyzed (Participants) | 10 | 12 | 10 | 9
  003 Week 24 Change from 002 Baseline | -11.6 (29.45) | 18.9 (41.08) | 29.2 (35.91) | 43.9 (43.72)

ADVERSE EVENTS:
Time Frame: Adverse events, including Serious Adverse Events (SAEs), and concomitant medications will be assessed at each study visit and recorded throughout the 24 week treatment period.
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/12 | 2/12
Other Adverse Events (participants affected / at risk) | 10/12 | 10/12 | 11/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level Group 1 (N=12) | Dose Level Group 2 (N=12) | Dose Level Group 3 (N=12) | Dose Level Group 4 (N=12)
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Testicular Torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level Group 1 (N=12) | Dose Level Group 2 (N=12) | Dose Level Group 3 (N=12) | Dose Level Group 4 (N=12)
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1
Excessive eye blinking (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 7 | 5 | 3
Thirst (General disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 2 | 1
Ear infection (Infections and infestations) | 1 | 1 | 1 | 1
Enterobiasis (Infections and infestations) | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 3
Otitis Media (Infections and infestations) | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 4 | 4 | 7 | 5
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Human Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood cortisol abnormal (Investigations) | 0 | 0 | 0 | 1
Urine output increased (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0
Abnormal behavior (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1
Stereotypy (Psychiatric disorders) | 1 | 0 | 0 | 0
Tic (Psychiatric disorders) | 1 | 0 | 0 | 0
Testicular Torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Uriticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02760277/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02760277/SAP_001.pdf